CLINICAL TRIAL: NCT04607785
Title: The Comparative Evaluation of Efficacy of 40% Miswak Mouthwash With 0.12% Chlorhexidine Mouthwash Among Gingivitis: A Blind Randomized Controlled Trial
Brief Title: Miswak Efficacy Compared With Chlorhexidine
Acronym: MiswakChlorx
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Al-Iraqia University (Other)
Responsible Party: Principal Investigator, Sumayah Al-Mahmood, Principal Investigator, Al-Iraqia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020DEN
Record Dates: First submitted 2020-10-09; First posted 2020-10-29 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Gingivitis
Keywords: Miswak; chlorhexidine; mouthwash; gingivitis; oral health
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Miswak mouthwash group (Active Comparator): Miswak sticks were bought from local markets, Baghdad, Iraq, washed with cold water and dried then crushed into powder. Later,7 grams of the miswak powder weighted and added to 350 ml of distilled water (D.W.) in a conical flask for 24 hours. Finally, the solution then filtered and stored in tightly closed bottles in a cool place.9
  Interventions: Drug: Miswak mouthwash group; Device: Chlorhexidine gluconate mouthwash
- Chlorhexidine mouthwash group (Other): 0.12% chlorhexidine gluconate mouthwash for seven days
  Interventions: Drug: Miswak mouthwash group; Device: Chlorhexidine gluconate mouthwash

INTERVENTIONS:
Drug: Miswak mouthwash group — Twice daily for seven days for two months
Device: Chlorhexidine gluconate mouthwash — Twice daily for seven days for two months
  Other Names: chlorhexidine gluconate Kin Gingival®

SUMMARY:
Gingivitis is a form of gum disease and is elicited by the accumulation of plaque on the tooth and the soft-tissue adjoining the tooth. Mouthwashes containing chemical or herbal substances are adjunctive tools in improving oral hygiene. Miswak mouthwash is a herbal mouthwash. Chlorhexidine mouthwash is the most efficient antimicrobial and antiplaque agent. The aim of the study is to assess the effectiveness of the miswak mouthwash with 0.12% chlorhexidine. This study was a blind randomized clinical trial.

Materials and Methods: A total of 60 patients aged (20-55) years old who attended the Periodontics Clinics at College of Dentistry, Al-Iraqia University were allocated for use the mouthwash either miswak mouthwash or 0.12% chlorhexidine gluconate Kin Gingival® (Laboratorios KIN, Spain) twice daily (once in the morning and one before bedtime) for seven days. Gingival, bleeding, and plaque indices were recorded at baseline and after 7 days of treatment.

DETAILED DESCRIPTION:
Gingivitis is the mildest form of gum disease and is elicited by the accumulation of plaque on the tooth and the soft-tissue adjoining the tooth. Accumulation of dental biofilm has been established as the initial cause of this disease. It is determined by redness of the gum margins, edema, bleeding upon brushing, and loss of periodontal attachment loss. Gingivitis exists in both acute and chronic forms. Acute gingivitis is identified as trauma, micro-organisms, and specific infections while chronic inflammation is related to bacterial biofilm which covers the gum and adjoining the teeth. Elimination and control of plaque are very important in the maintenance of periodontal health. Chlorhexidine mouthwash has is a tremendous effect when it is used as a mouthwash for a long time; therefore, the Food and Drug Administration (FDA) recommends limiting the use of chlorhexidine mouthwash up to 6 months to minimize or limit its side effects. Additionally, the World Health Organization (WHO) encouraged to consider the possible use of herb extracts and natural plants mouthwashes instead of chemical mouthwash just as miswak mouthwash. Miswak mouthwash is a herbal mouthwash that is available locally and culturally accepted. It is prepared from a plant called Salvadora persica which comes from a tree (Arak) that grows in Africa and west India.

ELIGIBILITY:
Inclusion Criteria:

* Adults with existence at least 20 natural teeth in the mouth
* Existence of lateral maxillary teeth
* Existence of central teeth
* Existence of mandibular teeth

Exclusion Criteria:

* Patients have no history of drug use
* Patients have no any disease relevant occurrence
* Pocket depth<3 mm
* Smokers
* Pregnancy

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Inflammation of gingiva | 2 months
  Change in Gingival index
Bleeding from gingiva | 2 months
  Change in index
Plaque in the gingiva | 2 months
  Change in index

CONTACTS AND LOCATIONS:
Locations (1):
- Dunia Wadeea Sabea, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
No need